CLINICAL TRIAL: NCT03209583
Title: ATrial Tachycardia PAcing Therapy in Congenital Heart
Acronym: AT-PATCH
Status: Recruiting | Type: Observational
Sponsor: Ian Law (Other)
Collaborators: Memorial Healthcare System (Other); Indiana University Health (Other); Mayo Clinic (Other); Rainbow Babies and Children's Hospital (Other); The Hospital for Sick Children (Other); University of Wisconsin, Madison (Other); University of California, Los Angeles (Other); University of Utah (Other); Norton Healthcare (Other); University of Michigan (Other); Vanderbilt University Medical Center (Other); Children's Hospital of Orange County (Other)
Responsible Party: Sponsor-Investigator, Ian Law, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201605847
Record Dates: First submitted 2017-06-07; First posted 2017-07-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-01

CONDITIONS: Atrial Arrhythmia; Atrial Tachycardia; Congenital Heart Disease; Pacemaker Re-Entrant Tachycardia
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Congenital Heart Disease: subjects have CHD and arrhythmias being treated with an implanted pacing device.
  Interventions: Device: Medtronic

INTERVENTIONS:
Device: Medtronic — Pacing is done by the implanted device after seeing how the electrical system is functioning giving energy when needed to maintain a stable state or rhythm

SUMMARY:
Congenital heart disease (CHD) affects approximately 1% of newborns in the US, with 25% of those affected having critical conditions requiring open heart surgery within one year of birth. Surgical and medical advances have allowed many patients to live beyond their fourth and fifth decades of life. Unfortunately, cardiac arrhythmias are a relatively common sequela due to cardiac anomalies and surgical scars in addition to residual volume and pressure load on the heart. Atrial arrhythmias, including sinus node dysfunction and intra-atrial re-entrant tachycardia (IART) are among the more common abnormalities found in adults with repaired CHD. The presence of IART significantly increases morbidity and mortality, and anti-arrhythmic medications have been shown to be a sub-optimal treatment strategy with the majority of patients requiring multi-drug therapy. Catheter ablation procedures remain a treatment option, but are less successful for some patient demographics. In the mid-1990's, pacemakers with atrial anti-tachycardia pacing (ATP) capabilities were developed, primarily for the management of atrial flutter and fibrillation in adults with structurally normal hearts. Given the need for pacemakers in the CHD population to manage sinus node dysfunction and atrioventricular node conduction block, the adoption of atrial anti-tachycardia pacemakers began to gain favor. However, there is limited data available comparing the safety and effectiveness of ATP therapy between various demographics of CHD patients. In the current study, the investigators aim to determine if ATP is an effective treatment strategy for IART, specifically within particular sub-populations of CHD patients. Additionally, investigators hope to delineate any significant differences in efficacy of ATP treatment between adult and pediatric congenital heart patients. The research team will accomplish our goals with a retrospective, multi-center study in which data is collected from existing electronic medical records and pacemaker interrogations. Following data collection, the investigators will employ statistical analyses to determine if certain CHD demographics are statistically significant predictors of ATP therapy outcomes.

The purpose of this prospective/retrospective study is to determine how effective atrial anti-tachycardia therapies are with the congenital heart patients who are known to have atrial arrhythmias. As this population ages, we know that arrhythmic burden increases and medications are increased or changed for symptomatic improvement.

Patients will be enrolled at the time of anti tachycardia device (ATD) placement or when device therapies are turned on. Patients will need a minimum of 5 years of clinical history prior to implantation and after implantation (unless patient is very young). Data will be collected both retrospectively and prospectively. The research team will consent patients at the time of clinical evaluations and scheduled follow-ups (usually 3 - 6 months). If therapy is effective, investigators will determine the specific programming which was successful. If therapy was ineffective, investigators will also determine if a change in programing was made and if this improved ATP efficacy. Investigators will also determine the arrhythmia burden. Cardioversion and medications before and after ATD implantation will be the key determinants of arrhythmia burden in this study.

DETAILED DESCRIPTION:
University of Iowa is moving to begin the multi-institutional portion of this study by asking for centers to assist with enrollment so that the investigators can meet our enrollment goal. The investigators wish to recruit a minimum of 250 subjects and will collect data for up to 300 subjects. The research team will move to a retrospective and prospective enrollment looking at how well ATP works in ATD therapy devices for patients who have CHD. No interventions will take place as this is a chart review and observational study.

ELIGIBILITY:
Inclusion Criteria:

* must have structural CHD, an atrial arrhythmia and an ATD implanted. ATP must be turned on.

Exclusion Criteria:

* Other arrhythmias substrates such as Long QT (LQT), hypertrophic Cardiomyopathy (HCM), Catecholaminergic polymorphic ventricular tachycardia (CPVT), Arrhythmogenic Right Ventricular Cardiomyopathy.(ARVC), Brugada & patients who undergo transplant, surgical maze, or ablation within 5 years of ATD implantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults with structural congenital heart disease, with documented atrial arrhythmia (IART, CHB, SND), and with an ATD which has therapies enabled. Patients will all be seen by providers at the University of Iowa Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
To measure any change in IART burden before and after ATD implantation. | 5 years at minimum
  The comparison will be how many times a cardioversion was needed and or how many times the device was able to or wasn't able to pace the heart out of the fast rate which could otherwise have been treated with a cardioversion. Data will be collected for a maximum of 5 years prior to implantation of an ATD and compared to a maximum of 5 years post implantation.

SECONDARY OUTCOMES:
Antiarrhythmic medication burden | 5 years at minimum
  IART is often treated with medication. The dose (mg/kg) for each medication needed to control arrhythmias before and after placement of and ATD will be reviewed.
Comparison of ATP protocols of RAMP vs. BURST + | 5 years at minimum.
  Once the ATD device is implanted there are two types of treatments the ATD is capable of implementing. The investigators will determine the % success rate for both of these treatment modalities for purposes of comparison.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (14):
  - University of California, Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County (CHOC), Orange, California
  - Memorial Healthcare System, Hollywood, Florida
  - Indiana University Health, Indianapolis, Indiana
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - Norton Healthcare, Louisville, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Madison, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Investigators are not sharing data with other researchers

REFERENCES:
- [Background] Kramer CC, Maldonado JR, Olson MD, Gingerich JC, Ochoa LA, Law IH. Safety and efficacy of atrial antitachycardia pacing in congenital heart disease. Heart Rhythm. 2018 Apr;15(4):543-547. doi: 10.1016/j.hrthm.2017.12.016. Epub 2017 Dec 12. PMID 29246827
- [Background] Kramer CC, Maldonado JR, Olson MD, Gingerich JC, Ochoa LA, Law IH. Atrial Antitachycardia Pacing in Complex Congenital Heart Disease: A Case Series. J Innov Card Rhythm Manag. 2018 Mar 15;9(3):3079-3083. doi: 10.19102/icrm.2018.090304. eCollection 2018 Mar. PMID 32477803